CLINICAL TRIAL: NCT02417090
Title: Metformin Therapy for Gestational Diabetes - Metabolic Late Effects on Child at 9 Years of Age
Brief Title: Late Metabolic Effects of Metformin Therapy in Gestational Diabetes
Acronym: DIARA2
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Harri Niinikoski, MD, Pediatric Endocrinologist, Professor of Nutrition in Medicine., Turku University Hospital
Other Study IDs: DIARA2
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational | interventions — Insulin; Insulin Lispro; Insulin Aspart; Metformin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Whole blood for DNA extraction
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Metformin therapy: 9-year-old children whose mothers used metformin for gestational diabetes
  Interventions: Drug: Metformin
- Insulin therapy: 9-year-old children whose mothers used insulin for gestational diabetes
  Interventions: Drug: Insulin

INTERVENTIONS:
Drug: Insulin — Pregnant women who used insulin to treat gestational diabetes
  Other Names: Humalog, Protaphane, Novorapid
  Groups: Insulin therapy
Drug: Metformin — Pregnant women who used metformin to treat gestational diabetes
  Other Names: Diformin retard
  Groups: Metformin therapy

SUMMARY:
Metformin in widely used as the treatment of gestational diabetes. However, it is not known whether exposure to metformin in utero has late metabolic effects on the child.

In this study the investigators investigate metabolism (oral glucose tolerance test, insulin, plasma lipoproteins, inflammation markers as well as body composition by DEXA (dual energy X-ray absorption) and MRI) in 9 year-old children whose mothers used either metformin of insulin during pregnancy.

DETAILED DESCRIPTION:
Gestational diabetes is usually managed with diet and insulin, if needed. However, oral metformin therapy has been also used to treat gestational diabetes and the short-term studies have shown that it is effective and also safe for the child. However, long-term studies of its effects are lacking.

Previously, several years ago, 217 pregnant women with gestational diabetes in Turku and 100 such women in Oulu, Finland, were randomised to either insulin or metformin therapy to treat gestational diabetes. In those studies, the metformin therapy proved to be safe in the short-term.

Now these children are 5-9 years old. In the present study these children (as well as their mothers) are investigated when the children are 9 years old. The aim is to study whether the metformin given during the pregnancy has any metabolic effects on the child at 9 years of age. To do this these families are contacted by mail and asked to participate into the study.

At 9 years of age, the following investigations will be made (after consent from the child and family): oral glucose tolerance test+insulin+c-peptide, plasma lipoproteins, adiponectin, PAI-1 (plasminogen activator inhibitor-1), IL-6 (interleukin-6), HS CRP (high-sensitivity C-reactive protein), p-metabolomics, DEXA, abdominal MRI, WISC IV (Wechsler intelligence scale for children IV)cognitive testing, BRIEF questionnaire, questionnaire about diet and health habits. The study subjects will also be clinically examined and measured and blood pressure will be taken.

All analyses are performed at the University hospital laboratory and radiology facilities using modern techniques. The amount of blood taken is limited and also radiation dose from DEXA is very small. The data are kept behind lock and key. Statistical analyses will be performed to study whether children exposed to metformin during pregnancy have any differences in their metabolism and well-being than those exposed to insulin. This study involves no new medical treatments to the study subjects.

ELIGIBILITY:
Inclusion Criteria:

* all children whose mothers used either metformin or insulin to treat gestational diabetes and were involved in the previous metformin study in Turku or Oulu, Finland

Exclusion Criteria:

* severe congenital malformations

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 9-year old children exposed to insulin or metformin in utero because their mothers had gestational diabetes
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2015-05; Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Metabolic late effects | 9 years
  To study possible late effects of gestational diabetes treated with metformin vs insulin

CONTACTS AND LOCATIONS:
Overall Officials: Harri J Niinikoski, MD, PhD, Principal Investigator — University of Turku

REFERENCES:
- [Background] Tertti K, Ekblad U, Koskinen P, Vahlberg T, Ronnemaa T. Metformin vs. insulin in gestational diabetes. A randomized study characterizing metformin patients needing additional insulin. Diabetes Obes Metab. 2013 Mar;15(3):246-51. doi: 10.1111/dom.12017. Epub 2012 Oct 24. PMID 23020608
- [Background] Ijas H, Vaarasmaki M, Morin-Papunen L, Keravuo R, Ebeling T, Saarela T, Raudaskoski T. Metformin should be considered in the treatment of gestational diabetes: a prospective randomised study. BJOG. 2011 Jun;118(7):880-5. doi: 10.1111/j.1471-0528.2010.02763.x. Epub 2010 Nov 18. PMID 21083860
- [Result] Tertti K, Ekblad U, Vahlberg T, Ronnemaa T. Comparison of metformin and insulin in the treatment of gestational diabetes: a retrospective, case-control study. Rev Diabet Stud. 2008 Summer;5(2):95-101. doi: 10.1900/RDS.2008.5.95. Epub 2008 Aug 10. PMID 18795211
- [Derived] Huhtala M, Ronnemaa T, Tertti K, Niinikoski H, Paavilainen E. Maternal and umbilical cord serum lipids in gestational diabetes predict offspring insulin secretion and resistance at the age of nine years. Metabolomics. 2025 Jun 22;21(4):87. doi: 10.1007/s11306-025-02281-9. PMID 40544417
- [Derived] Huhtala MS, Ronnemaa T, Paavilainen E, Niinikoski H, Pellonpera O, Juhila J, Tertti K. Prediction of pre-diabetes and type 2 diabetes nine years postpartum using serum metabolome in pregnant women with gestational diabetes requiring pharmacological treatment. J Diabetes Complications. 2023 Jul;37(7):108513. doi: 10.1016/j.jdiacomp.2023.108513. Epub 2023 May 26. PMID 37267720
- [Derived] Huhtala M, Nikkinen H, Paavilainen E, Niinikoski H, Vaarasmaki M, Loo BM, Ronnemaa T, Tertti K. Comparison of glucose metabolism and anthropometry in women with previous gestational diabetes treated with metformin vs. insulin: 9-year follow-up of two randomized trials. Acta Obstet Gynecol Scand. 2022 May;101(5):514-523. doi: 10.1111/aogs.14343. Epub 2022 Mar 11. PMID 35274295
- [Derived] Paavilainen E, Tertti K, Nikkinen H, Veijola R, Vaarasmaki M, Loo BM, Tossavainen P, Ronnemaa T, Niinikoski H. Metformin versus insulin therapy for gestational diabetes: Effects on offspring anthropometrics and metabolism at the age of 9 years: A follow-up study of two open-label, randomized controlled trials. Diabetes Obes Metab. 2022 Mar;24(3):402-410. doi: 10.1111/dom.14589. Epub 2021 Nov 24. PMID 34738701